CLINICAL TRIAL: NCT00770016
Title: Insulin Sensitivity and Metabolism Before and After Treatment in Patients With Hypothyroidism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no longer interested in doing the study
Sponsor: University of Aarhus (Other)
Collaborators: MR Research Center, Skejby Sygehus, Brendstrupgaardsvej 100, 8200 Aarhus N (Unknown)
Responsible Party: Jens Otto Lunde Jorgensen, Medical Department M, Aarhus University Hospital, Aarhus Sygehus, Norrebrogade 44, 8000 Aarhus C
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LM_HYPO_2008
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Hypothyroidism
Keywords: insulin sensitivity; Substrate metabolism; Fatty liver; intramyocellular lipid; intracellular signaling
MeSH Terms: conditions — Hypothyroidism; Insulin Resistance; Fatty Liver | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): the aim of the present study is to characterize the treatment related changes in insulin sensitivity, substrate metabolism and intrahepatic - intramyocellular lipids in 12 adult patients, recently diagnosed with hypothyroidism
  Interventions: Drug: Levothyroxin

INTERVENTIONS:
Drug: Levothyroxin — Dosage regulation will follow the local recommendations of treatment
  Other Names: Eltroxin (Levothyroxin, GlaxoSmithKline Pharma)

SUMMARY:
The aim of this study is to further characterize the treatment related changes in insulin sensitivity, substrate metabolism and intra hepatic- and intramyocellular lipid content in patients with hypothyroidism

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* must be of legal age and competent
* Age > 18 years
* presently diagnosed with hypothyroidism

Exclusion Criteria:

* alcohol consumption >21 units per week
* Malignant disease
* pregnancy
* magnetic implants or material in the body
* BMI > 30
* Heart disease (NYHA >2)
* Uncontrolled hypertension
* Manifest diabetes mellitus
* Changes in medication, with any influence on glucose metabolism, 2 months prior to and until the end of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2010-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
intracellular lipid content in liver and muscle | before and after 3 months treatment with growth hormone
intraabdominal lipid content | before and after treatment
insulin sensitivity | before and after treatment
substrate metabolism | before and after treatment
intracellular signaling in the basal state and during insulin stimulation | before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Medical department M (Endocrinology and Diabetes), Aarhus University Hospital, Aarhus Sygehus,, Aarhus, Denmark

REFERENCES:
- See also: Louise Møller — http://person.au.dk/da/louisem@dadlnet.dk/
- See also: (Danish Data Protection Agency) — http://www.datatilsynet.dk/english/